CLINICAL TRIAL: NCT06604273
Title: Unravelling Intestinal Fibrosis in Ulcerative Colitis
Acronym: INTERACT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dalia Lartey, Drs, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL85277.018; 2023-507907-73-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD); Fibroblast Activation Protein Inhibitor
Keywords: PET CT; FAPI; IBD; Ulcerative colitis; Filgotinib
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Half of the study participants will undergo PET CT imaging. Therefore, the interventional study model only applies to half of the study partcipants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 2 (Experimental): This group undergoes FAPi-PET CT imaging
  Interventions: Diagnostic Test: Fibroblast Activation Protein Inhibitor
- Group 1 (No Intervention): Does not undergo a FAPi scan

INTERVENTIONS:
Diagnostic Test: Fibroblast Activation Protein Inhibitor — PET CT imaging using the fibroblast activation protein inhibitor tracer
  Other Names: FAPi PET CT scan
  Arms: Group 2

SUMMARY:
The main objectives are: (i) to identify candidate fibrotic cellular pathways in UC patients treated with a JAK inhibitor filgotinib), and (ii) to detect and monitor in vivo fibrosis in UC patients using FAPi-PET/CT imaging

ELIGIBILITY:
Inclusion Criteria:

* Adults with confirmed diagnosis of UC - Group 1 criterion: ≥18 years of age regardless of gender
* Group 2 criterion: ≥30 years of age for males and ≥40 years of age for females
* Active disease confirmed by endoscopy (endoscopic Mayo score ≥ 2)
* Indication to start treatment with filgotinib

AND one of the following criteria:

* Active disease confirmed by intestinal ultrasound (BWT > 3 mm in at least one bowel segment and at least one other pathological IUS parameter) or
* Increased CRP (>5 mg/L) and/or fecal calprotectin levels (>250 mg/kg)

Exclusion Criteria:

* Pregnancy
* Unable to provide informed consent
* Colorectal carcinoma or high-grade dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Candidate fibrotic cellular pathways | From enrollment to end of study participation at 24 weeks
  Identification of candidate fibrotic cellular pathways using single cell pathway analysis and mucosal biopsies from UC patients before and at week 24 weeks after treatment initiation with filgotinib.

SECONDARY OUTCOMES:
68Ga-FAPi-PET/CT imaging feasibility | From enrollment to end of study participation at 24 weeks
  Feasilibility 68Ga-FAPi-PET/CT imaging as biomarker to monitor in vivo fibrosis in UC. By detection of in vivo intestinal fibrosis by means of measuring 68Ga-FAPi uptake, both visually as semi-quantitatively, in UC patients using FAPi-PET/CT imaging at baseline and 24 weeks after treatment initiation with filgotinib.
Correspondance 68Ga-FAPi uptake and STAT expression | From enrollment to end of study participation at 24 weeks
  To determine to what extent 68Ga-FAPi bowel uptake in UC patients corresponds to (phospohorylated and total) STAT gene and protein (i.e. down-stream JAK targets) expression
Correspondance 68Ga-FAPi uptake and clinical and endoscopic parameters | From enrollment to end of study participation at 24 weeks
  To determine to what extent 68Ga-FAPi bowel uptake in UC patients corresponds to clinical and endoscopic changes after 24 weeks of treatment with filgotinib

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lowenberg, MD PhD, Principal Investigator — Amsterdam University Medical Centers
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided